CLINICAL TRIAL: NCT04617769
Title: Effects of Antagonistic Actions in Response to Trauma Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Michael J. Telch, Professor, University of Texas at Austin
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00000113
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Post Traumatic Stress Disorder
Keywords: post traumatic stress disorder; PTSD; psychoeducation; exposure; trauma; combat; sexual assault; physical assault; motor vehicle accident
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Psychoeducation alone (PSYED) (Placebo Comparator): The participant will receive both PDF and video materials involving psychoeducational materials on trauma and safety behaviors.
  Interventions: Behavioral: Psychoeducation
- Psychoeducation followed by exposure (PSYED+EXP) (Active Comparator): The participant will receive both PDF and video materials involving psychoeducational materials on trauma and safety behaviors. The participant will then be instructed to start the trauma video clip exposures. There will be six 3-minute video exposure trials with an inter-trial interval of 2 minutes, during which participants will complete ratings of (a) peak subjective distress during the trauma-videoclip; (b) anticipated subjective distress for the next trial; and (c) level of confidence for coping with their own trauma memory should it become activated.
  Interventions: Behavioral: Psychoeducation; Behavioral: Exposure
- Psychoeducation & exposure/Antagonistic Actions (PSYED+EXP+AA) (Experimental): The participant will receive both PDF and video materials involving psychoeducational materials on trauma and safety behaviors. The participant will then be instructed to start the trauma video clip exposures. There will be six 3-minute video exposure trials with an inter-trial interval of 2 minutes, during which participants will complete ratings of (a) peak subjective distress during the trauma-videoclip; (b) anticipated subjective distress for the next trial; and (c) level of confidence for coping with their own trauma memory should it become activated. Antagonistic action strategies during exposure to the trauma-videoclips will include (a) adopting an open posture; (b) eating a palatable snack; (c) smiling; and (d) wishing on high levels of emotional distress (e.g., "come on distress hit me with your best shot"). The participant will engage in all of the four antagonistic actions for the six exposure trials.
  Interventions: Behavioral: Psychoeducation; Behavioral: Exposure

INTERVENTIONS:
Behavioral: Psychoeducation — psychoeducational materials on trauma and safety behaviors
Behavioral: Exposure — six 3-minute video exposure trials with an inter-trial interval of 2 minutes
  Arms: Psychoeducation & exposure/Antagonistic Actions (PSYED+EXP+AA); Psychoeducation followed by exposure (PSYED+EXP)

SUMMARY:
The overarching objective of this study is to investigate the use of antagonistic actions as a treatment augmentation strategy for enhancing emotional processing during exposure to trauma-relevant stimuli. To accomplish this, participants (N = 84) reporting exposure to a combat, sexual assault, physical assault, or motor vehicle accident Criterion A trauma will be randomized to one of three experimental conditions: (a) Psychoeducation alone (PSYED); (b) Psychoeducation followed by repeated exposure to trauma-videoclips (PSYED + EXP); or (c) Psychoeducation followed by repeated exposure to trauma-videoclips while engaging in antagonistic actions (PSYED + EXP + AA). Antagonistic action strategies during exposure to the trauma-videoclips will include (a) adopting an open posture; (b) eating a palatable snack; (c) smiling; and (d) wishing on high levels of emotional distress.

The investigators expect that (a) those randomized to receive psychoeducation alone will show less improvement relative to the two groups that receive psychoeducation plus repeated exposure to trauma-videoclips; (b) those receiving psychoeducation in combination with repeated exposure to trauma-videoclips while performing antagonistic actions will show significantly enhanced treatment outcome at the one-month follow-up relative to the other two treatment arms; (c) participants with greater PTSD symptom severity are likely to have a poorer treatment outcome to PSYED alone; (d) changes in trauma-related threat appraisals, coping self-efficacy, and safety behaviors will each independently mediate the effects of treatment; and (e) participants displaying reductions in their emotional reactivity are more likely to have a reduction in PTSD symptoms.

DETAILED DESCRIPTION:
Over 70% of Americans are exposed to trauma during their lifetime and approximately 5.6% will meet diagnostic criteria for posttraumatic stress disorder. Posttraumatic stress disorder (PTSD) can significantly interfere with social functioning, work, and increase one's risk for other physical and mental health problems. Trauma-focused psychotherapies for PTSD have been shown to outperform more traditional supportive psychotherapy or pharmacotherapy and have become the first line of treatment for PTSD. However, the impact of trauma-focused therapy such as Prolonged Exposure (PE) is reduced, due to high rates of attrition ranging from 38.5% to 50%. Thus, there is a clear need to develop treatments for PTSD that are more palatable.

Preliminary evidence suggests that exposure-based treatment may be enhanced by having patients engage in antagonistic actions (e.g., smiling, laughing, adopting an open posture, wishing on threatening outcomes) during exposure to the feared target. Prior research found that these actions increased the efficacy of exposure therapy among a sample of 88 patients with acrophobia. Specifically, participants were instructed to stand at the railing and look over the edge while shaking their head to induce dizziness, standing at the edge without holding onto the railing, or walking towards the railing with their eyes closed and hands behind their back. Participants in the antagonistic action exposure group exhibited a significantly greater reduction in peak fear over the course of the study compared to all other groups (89% reduction versus 54%). Although promising, augmenting exposure therapy with antagonistic actions has yet to be tested for enhancing exposure therapy for PTSD. For the present study, antagonistic actions will include (a) adopting an open posture; (b) eating a palatable snack; (c) smiling; and (d) wishing on high levels of emotional distress (e.g., "come on distress hit me with your best shot").

There is a gap in the literature on antagonistic actions related specifically to trauma exposure. By better understanding mechanisms underlying reactions to a trauma video clip and trauma symptom development, the investigators can begin to reduce the debilitating effects of psychopathology following exposure to traumatic events in the future.

The study is a 3 x 3 mixed model experimental design with treatment Condition as a three-level between-subjects factor and assessment period (baseline vs posttreatment vs follow-up) as a three-level within subjects factor. Participants (N = 84) reporting exposure to a combat, sexual assault, physical assault, or motor vehicle accident Criterion A trauma will complete a battery of baseline trauma-related symptom measures followed by a trauma memory provocation involving watching a brief trauma-relevant videoclip, during which behavioral and subjective indices of emotional reactivity will be collected. Participants will be stratified based on their trauma symptom severity (PCL-5) and trauma type (LEC-5) and then randomized to one of three conditions: (a) Psychoeducation alone (PSYED); (b) Psychoeducation followed by repeated exposure to trauma-videoclips (PSYED + EXP); or (c) Psychoeducation followed by repeated exposure to trauma-videoclips while engaging in antagonistic actions (PSYED + EXP + AA). Antagonistic action strategies during exposure to the trauma-videoclips will include (a) adopting an open posture; (b) eating a palatable snack; (c) smiling; and (d) wishing on high levels of emotional distress (e.g., "come on distress hit me with your best shot").

Participants randomized to the two trauma videoclip exposure arms will receive six 3-minute video exposure trials with an inter-trial interval of 2 minutes, during which participants will complete ratings of (a) peak subjective distress during the trauma-videoclip; (b) anticipated subjective distress for the next trial; and (c) level of confidence for coping with their own trauma memory.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 60
2. Speaks English fluently
3. Identify either an assault, motor vehicle accident, or combat index trauma on the LEC-5
4. Access to the internet
5. Willingness to provide signed informed consent
6. Willingness to refrain from all non-study trauma-focused treatment during the study period

Exclusion Criteria:

1. History of a suicide attempt within the past 6 months
2. Not displaying emotional reactivity during the baseline trauma video clip provocation challenge

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder Scale (PCL-5) | One month follow-up assessment
  Change from baseline in patient-rated PTSD severity. The subjective 20-item self-report measure assesses the 20 DSM-5 symptoms of PTSD, and is rated on a 5-point Likert-style scale (0 = not at all to 4 = extremely) with a maximum score of 80 indicating extreme distress from PTSD symptoms.

SECONDARY OUTCOMES:
Subjective Units of Distress (SUDs) | One month follow-up assessment
  Change from baseline in patient-rated subjective and behavioral indices of emotional reactivity to a new trauma-relevant videoclip, where higher scores indicate more distress.
PTSD-Relevant Threat Appraisals (PTA) | One month follow-up assessment
  Change from baseline in patient-rated PTSD-relevant threat appraisals, where higher score indicate greater perceived threat towards the trauma video clip.
Coping Self-Efficacy (CSE-T-SF) | One month follow-up assessment
  Change from baseline in patient-rated coping self-efficacy, where higher scores indicate greater perceptions of trauma-related self-efficacy coping
PTSD Safety Behavior Inventory (PSBI) | One month follow-up assessment
  Change from baseline in patient-rated trauma-related safety behaviors, where higher scores indicate greater usage of PTSD-related safety behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frans O, Rimmo PA, Aberg L, Fredrikson M. Trauma exposure and post-traumatic stress disorder in the general population. Acta Psychiatr Scand. 2005 Apr;111(4):291-9. doi: 10.1111/j.1600-0447.2004.00463.x. PMID 15740465
- [Background] Committee on the Assessment of Ongoing Efforts in the Treatment of Posttraumatic Stress Disorder; Board on the Health of Select Populations; Institute of Medicine. Treatment for Posttraumatic Stress Disorder in Military and Veteran Populations: Final Assessment. Washington (DC): National Academies Press (US); 2014 Jun 17. Available from http://www.ncbi.nlm.nih.gov/books/NBK224878/ PMID 25077185
- [Background] Kehle-Forbes SM, Meis LA, Spoont MR, Polusny MA. Treatment initiation and dropout from prolonged exposure and cognitive processing therapy in a VA outpatient clinic. Psychol Trauma. 2016 Jan;8(1):107-114. doi: 10.1037/tra0000065. Epub 2015 Jun 29. PMID 26121175
- [Background] Kessler RC. Posttraumatic stress disorder: the burden to the individual and to society. J Clin Psychiatry. 2000;61 Suppl 5:4-12; discussion 13-4. PMID 10761674
- [Background] McDevitt-Murphy ME, Williams JL, Bracken KL, Fields JA, Monahan CJ, Murphy JG. PTSD symptoms, hazardous drinking, and health functioning among U.S.OEF and OIF veterans presenting to primary care. J Trauma Stress. 2010 Feb;23(1):108-11. doi: 10.1002/jts.20482. PMID 20104586
- [Background] Perkonigg A, Kessler RC, Storz S, Wittchen H -U. Traumatic events and post-traumatic stress disorder in the community: prevalence, risk factors and comorbidity. Acta Psychiatr Scand. 2000 Jan;101(1):46-59. doi: 10.1034/j.1600-0447.2000.101001046.x. PMID 10674950
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Schottenbauer MA, Glass CR, Arnkoff DB, Tendick V, Gray SH. Nonresponse and dropout rates in outcome studies on PTSD: review and methodological considerations. Psychiatry. 2008 Summer;71(2):134-68. doi: 10.1521/psyc.2008.71.2.134. PMID 18573035
- [Background] Shalev AY, Gevonden M, Ratanatharathorn A, Laska E, van der Mei WF, Qi W, Lowe S, Lai BS, Bryant RA, Delahanty D, Matsuoka YJ, Olff M, Schnyder U, Seedat S, deRoon-Cassini TA, Kessler RC, Koenen KC; International Consortium to Predict PTSD. Estimating the risk of PTSD in recent trauma survivors: results of the International Consortium to Predict PTSD (ICPP). World Psychiatry. 2019 Feb;18(1):77-87. doi: 10.1002/wps.20608. PMID 30600620
- [Background] Wolitzky KB, Telch MJ. Augmenting in vivo exposure with fear antagonistic actions: a preliminary test. Behav Ther. 2009 Mar;40(1):57-71. doi: 10.1016/j.beth.2007.12.006. Epub 2008 Jul 2. PMID 19187817